CLINICAL TRIAL: NCT00301600
Title: Mycophenolate Mofetil Versus Intravenous Cyclophosphamide Pulses in the Treatment of Crescentic IgA Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine, Nanjing University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NJCT-0606
Record Dates: First submitted 2006-03-10; First posted 2006-03-13 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2008-07

CONDITIONS: IGA Nephropathy
Keywords: Crescentic IgA nephropathy; Mycophenolate mofetil; Cyclophosphamide; treatment
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mycophenolate mofeti (Active Comparator)
  Interventions: Drug: Mycophenolate mofetil

INTERVENTIONS:
Drug: Mycophenolate mofetil — MMF,1.0g/d
  Other Names: MMF,cellcept

SUMMARY:
A single-center random parallel study to compare the efficacy and safety of Mycophenolate mofetil versus intravenous Cyclophosphamide pulses in the treatment of crescentic IgA nephropathy

DETAILED DESCRIPTION:
IgA nephropathy is an immune-complex glomerulopathy that can result in capillary necrosis or extracapillary proliferation (crescents). Several studies have documented a higher incidence of hypertension and nephritic-range proteinuria in patients with the crescentic form of IgA nephropathy, suggesting that patients with this variant of the disease may have a worse prognosis. Some studies have shown that treatment with steroids and cyclophosphamide had efficacy on reducing proteinuria and preserving renal function by healing vasculitic lesions, therefore preventing the progression of glomerular sclerosis. Recent studies have also shown that mycophenolate mofetil is effective in the treatment of lupus nephritis with vasculitic lesion and small vasculitis with renal involvement. We will conduct a single-center prospective open-labeled clinical trial of 40 patients with crescentic IgA nephropathy and treat them randomly with pulse intravenous cyclophosphamide or oral mycophenolate mofetil. After 12 months of treatment, we will assess the efficacy, safety, tolerability and relapse of mycophenolate mofetil compared with cyclophosphamide in the treatment of crescentic IgA nephropathy.

ELIGIBILITY:
Inclusion Criteria:

Patient with a diagnosis of IgAN without deposition of C4 and C1q, age 10-70y, sex free

1. Gross hematuria or an active urine sediment
2. Segmental necrotizing lesion of the capillary wall
3. Cellular or fibrocellular crescents ≥ 10%
4. Fibrinoid degeneration of small vessels
5. Fibrin positive Three or more items, with provision of criteria informed consent

Exclusion Criteria:

1. More than four-week treatment with cytotoxic drug, such as CTX, CsA and MMF, prior to enrollment
2. Immune deficiency
3. Serum creatinine ≥ 5.0mg/dl
4. Previous malignancy
5. Pregnancy
6. Hepatitis
7. Diabetic mellitus or obesity
8. Severe infection or CVS complications
9. Henoch-Schonlein purpura nephritis, systemic vasculitis, SLE

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2003-01; Primary Completion 2005-05 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy and safety of Mycophenolate mofetil versus intravenous Cyclophosphamide pulses in the treatment of crescentic IgA nephropathy | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lei-Shi Li, M.D., Study Chair — Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine
Locations (1):
- Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Alladin A, Hahn D, Hodson EM, Ravani P, Pfister K, Quinn RR, Samuel SM. Immunosuppressive therapy for IgA nephropathy in children. Cochrane Database Syst Rev. 2024 Jun 12;6(6):CD015060. doi: 10.1002/14651858.CD015060.pub2. PMID 38864363